CLINICAL TRIAL: NCT06976775
Title: Comparative Analysis Between Two Oral Immunotherapy Schemes in Cow´s Milk and/or Hen´s Egg Allergic Children to Improve Treatment Efficiency and Identify Response Biomarkers. CompITO Study
Brief Title: Comparison Between a Rush and a Conventional Oral Immunotherapy Protocol to Treat Cow's Milk and Hen´s Egg Allergy. CompITO Study
Acronym: compITO
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pablo Rodríguez del Rio (Other)
Responsible Party: Sponsor-Investigator, Pablo Rodríguez del Rio, Sponsor-Investigator, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Organization: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: compITO
Record Dates: First submitted 2025-04-18; First posted 2025-05-16 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Food Allergy in Children; Milk Allergy; Egg Allergy
Keywords: Food immunotherapy; Allergy; Milk; Egg; Oral immunotherapy; Anaphylaxis; Mast cell activation test; Saliva; Blood; IgE; Food allergy; Sensitization; Children; Pediatric
MeSH Terms: conditions — Milk Hypersensitivity; Egg Hypersensitivity; Hypersensitivity; Anaphylaxis; Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rush protocol (Experimental): Milk and egg allergic children undergoing OIT following a Rush regimen
  Interventions: Biological: "Rush" regimen
- Conventional protocol (Active Comparator): Milk and egg allergic children undergoing OIT following a Conventional regimen
  Interventions: Biological: "Conventional" regimen

INTERVENTIONS:
Biological: "Rush" regimen — The "rush" regimen consists of the administration of several incremental doses daily, every day, over the first week of the Induction Phase (Part 1)
  Arms: Rush protocol
Biological: "Conventional" regimen — The "conventional" regimen consists of the administration of only one incremental dose every 2 weeks, throughout all the Induction Phase (Part 1)
  Arms: Conventional protocol

SUMMARY:
This study investigates the efficacy and safety of two different OIT schemes to treat milk and egg allergic children

DETAILED DESCRIPTION:
Food immunotherapy, especially oral immunotherapy (OIT), is now a standard treatment option for patients allergic to cow´s milk, hen´s egg or peanuts. While peanut OIT has drawn considerable attention from the scientific community, milk and hen´s egg OIT still remain as the most common immunotherapy administered in daily routine. Optimization of these treatments is a priority to offer to a wider number of candidates a more efficient and safe way of treatment.

A Phase II/III randomized clinical trial enrolling a total of 40 patients with non-severe food allergies (20 cow's milk allergic children and 20 hen's egg allergic children) to assess the safety and efficacy of a rush/rapid versus a conventional OIT protocol.

Schemes are comparable in terms of the number of doses, the relative increment between doses and the final amount of protein, with one exception: the "rush" regimen includes several doses given the same day over the first week of treatment while in the "conventional" regimen Induction Phase is based upon single doses given every 2 weeks.

There are two different parts in the study, during Induction Phase (Part 1, 1 week up to 7 months), participants in both groups will receive incremental doses of milk/egg, depending on their allergy, until they tolerate 6600 mg or 4680mg of milk or egg protein respectively. The occurrence of adverse events in both groups will result in dose adjustments and delay in completion Induction Phase. During Maintenance Phase (Part 2), patients will ingest the same dose (daily for milk and every 48h for egg) until the end of study, that will last for a total duration of 7 months.

The study features a dual primary outcome. Safety and efficacy variables are primary outcomes, and parents and patient-reported food allergy-related quality of life (HRQoL) are secondary outcomes, as well as burden of treatment and immunological changes. Molecular changes underlying OIT will be studied, and biomarkers of safety and efficacy will be sought

ELIGIBILITY:
Inclusion Criteria:

* Patients 6 to 16 years old
* sIgE levels to milk 0.35 to 35kUA/L for milk allergic subjects and egg 0.35 to 35kUA/L for egg allergic subjects
* Entry DBPCFC discrete milk eliciting dose (ED)≥ 22.2mg of milk protein and discrete egg ED≥18.5mg of egg protein, that are the population-based reference values for the ED20
* Having a mild to moderate food allergy severity per DEFASE score (<13 points)

Exclusion Criteria:

* sIgE levels to milk >35kUA/L for milk allergic subjects and egg > 35kUA/L for milk allergic subjects
* Entry DBPCFC discrete milk ED<22.2mg of milk protein or discrete egg ED<18.5mg of egg protein
* Entry DBPCFC discrete ED for milk>2112mg of milk protein (cumulative amount of 4193,7mg of milk protein) and egg discrete ED>1560mg of egg protein (cumulative amount of 3110.8mg of egg protein)
* Having severe food allergy per DEFASE score (≥13 points)
* Other exclusion criteria: uncontrolled asthma, FEV1<70%, severe atopic dermatitis, Eosinophilic Esophagitis, non-IgE mediated allergy, having started SCIT 3 months before, or SLIT one week before. Pregnancy

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events with an oFASS5 severity ≥2 occurred until Induction Phase (Part 1) completion at the hospital setting per subject in both groups, rush vs conventional | Throughout the Induction Phase (Part 1), 1 week up to 7 months
Proportion of subjects completing the Induction Phase (Part 1) in both groups (rush vs conventional) at the end of study (7 months of treatment) | End of study (7 months of treatment)

SECONDARY OUTCOMES:
Number of adverse events with an oFASS5 severity ≥2 reported until Induction Phase (Part 1) completion at home and hospital setting per subject in both groups, rush vs conventional | Throughout the Induction Phase (Part 1), 1 week up to 7 months
Number of anaphylaxis events reported until Induction Phase (Part 1) completion at home and hospital setting per subject in both groups, rush vs conventional | Throughout the Induction Phase (Part 1), 1 week up to 7 months
Comparison of the median threshold change between baseline double blind placebo-controlled food challenge (DBPCFC) and maximum tolerated dose (mg of protein) between rush and conventional protocol subjects at the end of the study (7 months of treatment) | End of study (7 months of treatment)
Comparison of the median number of days needed in both groups, rush vs conventional, to complete the Induction Phase (Part 1) in subjects accomplishing this outcome | Throughout the Induction Phase (Part 1), 1 week up to 7 months
Comparison of the median Food Allergy Quality of Life Questionnaire, Parental Form (FAQLQ-PF) score change in patients undergoing rush vs conventional protocols between baseline and end of study (7 months of treatment). | End of study (7 months of treatment)
  FAQLQ-PF values range from 0 to 6, with higher scores representing more QoL impairment
Comparison of the median burden of treatment score in patients undergoing rush vs conventional protocols at the end of study (7 months of treatment) | End of study (7 months of treatment)
  Burden of treatment evaluation will be carried out applying a new tool in current development, where values range from 0 to 6, and with higher scores representing a more burdensome treatment
Comparison of the median sIgE levels (kU/L) to milk or egg proteins in patients undergoing rush vs conventional protocols at baseline and at end of study (7 months of treatment) | End of study (7 months of treatment)
Comparison of the median SPT (mm) wheal size to milk or egg proteins in patients undergoing rush vs conventional protocols at baseline and at end of study (7 months of treatment) | End of study (7 months of treatment)
Comparison of the median sIgG4 (mg/L) levels to milk or egg proteins in patients undergoing rush vs conventional protocols at baseline and at end of study (7 months of treatment) | End of study (7 months of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Pablo Rodriguez del Río, MD, PhD, Principal Investigator — Hospital Infantil Niño Jesús, Instituto de Investigación La Princesa
Locations (1):
- Hospital Infantil Universitario Niño Jesús. Avenida de Menéndez Pelayo, número 65, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No